CLINICAL TRIAL: NCT01827748
Title: Evaluation of a Surgical Microscope Mounted Autorefractor When Used on Patients Lying in a Supine Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adventus Technology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: FA120928
Record Dates: First submitted 2013-03-29; First posted 2013-04-10 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Refractive Error
Keywords: Autorefractor
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intraoperative Autorefractor IAR-1 (Experimental): This is a auto refractor mounted on an operating microscope.
  Interventions: Device: Intraoperative Autorefractor IAR-1
- Hartmann-Shack Auto Refractor (Active Comparator): The Hartmann-Shack type auto refractor used with the subject sitting upright in front of the instrument.
  Interventions: Device: Hartmann-Shack Auto Refractor

INTERVENTIONS:
Device: Intraoperative Autorefractor IAR-1 — This is an auto-refractor mounted on an operating microscope and used with the subject in a supine position
  Arms: Intraoperative Autorefractor IAR-1
Device: Hartmann-Shack Auto Refractor — Standard auto-refractor used with subject sitting upright in front of the instrument.
  Arms: Hartmann-Shack Auto Refractor

SUMMARY:
The purpose of this study is to evaluate the accuracy and repeatability of an individually validated prototype autorefractor designed to be mounted on a surgical microscope.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the accuracy and repeatability of an individually validated prototype autorefractor designed to be mounted on a surgical microscope. The goal is to evaluate 20 subjects with both the investigational instrument followed by a commercially available instrument.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age as of the date of evaluation for the study.
2. Have:

   1. Read the Informed Consent
   2. been given an explanation of the Informed Consent
   3. indicated understanding of the Informed Consent
   4. signed the Informed Consent document.
3. Be willing and able to adhere to the instructions set forth in this protocol and able to participate in all scheduled evaluations.
4. Be in good general health, based on his/her knowledge.
5. Have a refractive error within the range of -10.00 to +30.00 Diopter sphere and up to 5.00 Diopter of refractive cylinder .
6. Have manifest refraction (BCVA) Snellen visual acuities (VA) equal to or better than 20/25 in each eye. -

Exclusion Criteria:

Subjects may not be enrolled in this study if any of the following apply: The subject is/has:

1. Allergy to Tropicamide or a previous adverse reaction to Tropicamide.
2. Poor personal hygiene as observed by the investigational site personnel.
3. Strabismus
4. Currently pregnant (to the best of the subject's knowledge) or is lactating.
5. Previous refractive surgery or current or previous orthokeratology treatment.
6. Aphakic or pseudophakic or has cataracts that interfere with visual acuity.
7. Ocular or systemic disease such as, but not limited to: anterior uveitis or iritis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, sclerodermia, keratoconus or type II diabetes.
8. The need for topical ocular medications or any medication which might interfere with the study evaluations.
9. The presence of clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
10. Slit lamp findings, including but not limited to:

Pathological dry eye or associated dry eye symptoms with decreased tear levels and punctuate staining > Grade 2 Pterygium Corneal scars within the visual axis Neovascularization or ghost vessels > 1.0 mm in from the limbus Giant papillary conjunctivitis (GPC) of > Grade 2 Anterior uveitis or iritis Seborrheic eczema, seborrheic conjunctivitis or blepharitis

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the accuracy and repeatability of the Test device compared to the Control | 1 Hour
  Comparative auto refractor device measurement variation is defined as +/-0.25 Diopters

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Berdy, MD, Principal Investigator
Locations (1):
- Ophthalmology Associates, St Louis, Missouri, United States